CLINICAL TRIAL: NCT01542307
Title: Normobaric Oxygen (NBO) Therapy in Acute Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Aneesh B. Singhal, MD, Associate Professor of Neurology, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009P000380; 2009P000380 (Other: PHRC)
Record Dates: First submitted 2012-02-21; First posted 2012-03-02 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: Migraine
Keywords: migraine; oxygen therapy
MeSH Terms: conditions — Migraine Disorders | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxygen (Experimental): Oxygen is inhaled for 30 minutes during migraine attack
  Interventions: Biological: Oxygen
- Room Air (Placebo Comparator): Medical air inhaled for 30 minutes during migraine attack
  Interventions: Biological: Room air

INTERVENTIONS:
Biological: Oxygen — Oxygen is inhaled for 30 minutes during migraine attack
  Arms: Oxygen
Biological: Room air — Placebo
  Arms: Room Air

SUMMARY:
This is a pilot study investigating the therapeutic potential of breathing 100% oxygen in acute migraine headache.

DETAILED DESCRIPTION:
A total of 40 adult subjects will be enrolled, male and female. Subjects will be consented to inhale either Normobaric Oxygen (NBO) or Room air for 30 minutes at the start of their migraine attacks. Outcomes will be assessed during and after gas treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects with frequent migraine (at least 1 attack per month)

Exclusion Criteria:

* Secondary (non-migraine) headache
* Chronic obstructive pulmonary disease
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aneesh B Singhal, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Singhal AB, Maas MB, Goldstein JN, Mills BB, Chen DW, Ayata C, Kacmarek RM, Topcuoglu MA. High-flow oxygen therapy for treatment of acute migraine: A randomized crossover trial. Cephalalgia. 2017 Jul;37(8):730-736. doi: 10.1177/0333102416651453. Epub 2016 May 20. PMID 27206964

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 22 subjects enrolled
Pre-assignment Details: 22 subjects enrolled - each subject generated data for one or more migraine attacks.
Units Other Than Participants: migraine attacks
Groups:
- Oxygen-treated Migraine Attacks: Oxygen is inhaled for 30 minutes during a migraine attack
- Medical Air-treated Migraine Attacks: Medical air is inhaled for 30 minutes during a migraine attack
Period: Overall Study
Arm/Group | Oxygen-treated Migraine Attacks | Medical Air-treated Migraine Attacks
Started | 22; 33 migraine attacks (Each subject inhaled Oxygen for 30 minutes in blinded fashion for 2 of the 4 migraine attacks) | 22; 31 migraine attacks (Each subject inhaled Medical Air for 30 minutes in blinded fashion for 2 of the 4 migraine attacks)
Completed | 22; 33 migraine attacks | 22; 30 migraine attacks
Not Completed | 0; 0 migraine attacks | 0; 1 migraine attacks

BASELINE CHARACTERISTICS:
Population: Enrolled subjects
Groups:
- Enrolled Subjects: Oxygen or Medical Air is inhaled in random order for 30 minutes during each migraine attack (total 4 attacks)
Arm/Group | Enrolled Subjects
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 20
  Non-Caucasian | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22
Migraine [Count of Participants; unit: Participants]
  Migraine w Aura | 7
  Migraine without Aura | 15
Employment [Count of Participants; unit: Participants]
  Employed Full Time | 17
  Not Employed Full Time | 5
Education Level [Count of Participants; unit: Participants]
  College or higher | 20
  School or lower | 2
Marital status [Count of Participants; unit: Participants]
  Married | 10
  Single | 12
Smoking Status [Count of Participants; unit: Participants]
  Prior smoker | 2
  Non-smoker | 20
Family history of migraine [Count of Participants; unit: Participants]
  Present | 13
  Absent | 9
Vascular risk factors (eg. hypertension) [Count of Participants; unit: Participants]
  Present | 2
  Absent | 20
One or more lifetime ED visits [Count of Participants; unit: Participants]
  Yes | 17
  None | 5
One or more ED visits in prior year [Count of Participants; unit: Participants]
  Visited | 11
  Not visited | 11
Triptans for acute migraine [Count of Participants; unit: Participants]
  Using | 18
  Not Using | 4
NSAIDs/acetaminophen for acute migraine [Count of Participants; unit: Participants]
  Using | 22
  Not Using | 0
Opioids for acute migraine [Count of Participants; unit: Participants]
  Using | 6
  Not Using | 16
Anti-seizure meds for migraine prevention [Count of Participants; unit: Participants]
  Using | 10
  Not Using | 12
Beta-blockers for migraine prevention [Count of Participants; unit: Participants]
  Using | 8
  Not Using | 14
Using botulinum toxin for migraine prevention [Count of Participants; unit: Participants]
  Using | 4
  Not Using | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Scores From 0-30 Minutes on a Visual Analog Scale (VAS)
Description: The mean change in VAS pain scores from 0 minutes to 30 minutes was selected as the primary outcome measure.
  The VAS scale has a range from 0-10 with higher scores indicating greater severity of symptoms.
Time Frame: From baseline (0 minutes) to 30 mins
Population: Number of migraine attacks treated with Oxygen or Medical Air
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Migraine attacks
Arm/Group | Oxygen | Room Air
Number analyzed (Participants) | 22 | 22
Number analyzed (Migraine attacks) | 33 | 31
units on a scale | 1.38 (1.42) | 1.22 (1.61)
Statistical Analysis 1: Comparison: Oxygen vs Room Air; Test type: Superiority or Other; p = 0.674, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in Pain Score From 0-15 Minutes on the Visual Analogue Scale (VAS)
Description: The mean change in VAS pain scores from 0 minutes to 15 minutes was selected as a secondary outcome measure.
  The VAS scale has a range from 0-10 with higher scores indicating greater severity of symptoms.
Time Frame: Baseline (0 minutes) to 15 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Migraine attacks
Arm/Group | Oxygen | Room Air
Number analyzed (Participants) | 22 | 22
Number analyzed (Migraine attacks) | 33 | 31
units on a scale | 0.77 (1.09) | 0.44 (0.92)
Statistical Analysis 1: Comparison: Oxygen vs Room Air; Test type: Superiority or Other; p = 0.18, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Pain Score From 0-60 Minutes on the Visual Analogue Scale (VAS)
Description: The mean change in VAS pain scores from 0 minutes to 60 minutes was selected as a secondary outcome measure.
  The VAS scale has a range from 0-10 with higher scores indicating greater severity of symptoms.
Time Frame: Baseline (0 minutes) to 60 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Migraine attacks
Arm/Group | Oxygen | Room Air
Number analyzed (Participants) | 22 | 22
Number analyzed (Migraine attacks) | 33 | 31
units on a scale | 2.05 (2.23) | 1.57 (1.94)
Statistical Analysis 1: Comparison: Oxygen vs Room Air; Test type: Superiority or Other; p = 0.38, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Final Pain Severity Score 0-1 on the Visual Analogue Scale (VAS)
Description: The percentage of migraine attacks with the final (60 minute) VAS pain score 0-1 was selected as a secondary outcome measure.
  The VAS scale has a range from 0-10 with higher scores indicating greater severity of symptoms.
Time Frame: 60 minutes
Measure: Number; unit: percentage of attacks
Units Other Than Participants: Migraine attacks
Arm/Group | Oxygen | Room Air
Number analyzed (Participants) | 22 | 22
Number analyzed (Migraine attacks) | 33 | 31
percentage of attacks | 24 | 6
Statistical Analysis 1: Comparison: Oxygen vs Room Air; Test type: Superiority or Other; p = 0.05, Fisher Exact

5. Secondary Outcome: Final Pain Score 0-1 or Score Improved 3 or More Points on the Visual Analogue Scale (VAS)
Description: The percentage of migraine attacks with the final (60 minute) VAS pain score either 0-1, or a 3-point improvement from baseline, was selected as a secondary outcome measure.
  The VAS scale has a range from 0-10 with higher scores indicating greater severity of symptoms.
Time Frame: 60 minutes
Measure: Number; unit: percentage of attacks
Units Other Than Participants: Migraine attacks
Arm/Group | Oxygen | Room Air
Number analyzed (Participants) | 22 | 22
Number analyzed (Migraine attacks) | 33 | 31
percentage of attacks | 45 | 23
Statistical Analysis 1: Comparison: Oxygen vs Room Air; Test type: Superiority or Other; p = 0.05, Fisher Exact

6. Secondary Outcome: Final Visual Symptom Score 0-1 on the Visual Analog Scale (VAS)
Description: The percentage of migraine attacks with the final (60 minute) VAS visual symptom score 0-1 was selected as a secondary outcome measure.
  The VAS scale has a range from 0-10 with higher scores indicating greater severity of symptoms.
Time Frame: 60 minutes
Measure: Number; unit: percentage of attacks
Units Other Than Participants: Migraine attacks
Arm/Group | Oxygen | Room Air
Number analyzed (Participants) | 22 | 22
Number analyzed (Migraine attacks) | 33 | 31
percentage of attacks | 36 | 6
Statistical Analysis 1: Comparison: Oxygen vs Room Air; Test type: Superiority or Other; p = 0.004, Fisher Exact

7. Secondary Outcome: Final Nausea Score 0-1 on the Visual Analog Scale (VAS)
Description: The percentage of migraine attacks with the final (60 minute) VAS nausea score 0-1 was selected as a secondary outcome measure.
  The VAS scale has a range from 0-10 with higher scores indicating greater severity of symptoms.
Time Frame: 60 minutes
Measure: Number; unit: percentage of attacks
Units Other Than Participants: Migraine attacks
Arm/Group | Oxygen | Room Air
Number analyzed (Participants) | 22 | 22
Number analyzed (Migraine attacks) | 33 | 31
percentage of attacks | 64 | 65
Statistical Analysis 1: Comparison: Oxygen vs Room Air; Test type: Superiority or Other; p = 1.00, Fisher Exact

8. Other Pre Specified Outcome: Post-gas Therapy Medication Use
Description: The percentage of migraine attacks requiring the use of one or more anti-migraine medications after the period of gas inhalation, was selected as a secondary outcome measure.
Time Frame: 60 minutes
Measure: Number; unit: percentage of attacks
Units Other Than Participants: Migraine attacks
Arm/Group | Oxygen | Room Air
Number analyzed (Participants) | 22 | 22
Number analyzed (Migraine attacks) | 33 | 31
percentage of attacks | 36 | 52
Statistical Analysis 1: Comparison: Oxygen vs Room Air; Test type: Superiority or Other; p = 0.16, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of enrollment and until a maximum of 4 migraine attacks were treated with gas inhalation and study equipment returned to the study team.
Description: Specific adverse events ('events of interest') were monitored around the time of each migraine attack (individual subjects had 1-4 migraine attacks each).
Arm/Group | Oxygen | Room Air
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 2/22 | 2/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxygen (N=22) | Room Air (N=22)
Dry Mouth (General disorders) | 1 (1) | 0 (0)
Tingling (Nervous system disorders) | 1 (1) | 0 (0)
Significant worsening of migraine headache (Nervous system disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No